CLINICAL TRIAL: NCT06350747
Title: The Effectiveness of Online and Face-to-Face Laughter Yoga on Nurses' Perceived Stress, Sleep Quality, and Burnout: A Three-Group Randomized Controlled Trial
Brief Title: The Effect of Laughter Yoga on Nurses' Perceived Stress, Sleep Quality, and Burnout Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Celal Bayar University (Other)
Responsible Party: Principal Investigator, Özge Topsakal, Principal Investigator, Celal Bayar University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CelalBayarU-SBF-OT-02
Record Dates: First submitted 2024-03-30; First posted 2024-04-05 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Healthy Participants
Keywords: burnout level; laughter yoga; nurses; stress; sleep quality
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: pretest-posttest with control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control Group (Other): Participants in this group did not receive any intervention during the study period. They only completed the pre- and post-intervention assessments. After study completion, they were offered a single optional laughter yoga session.
  Interventions: Other: control group
- Face-to-Face Laughter Yoga Group (Experimental): Participants in this group attended four sessions of laughter yoga conducted in person by certified instructors. Sessions lasted approximately 40 minutes and were held twice a week for two weeks in groups of 5-6 nurses.This intervention included hand clapping and warm-up exercises, deep breathing, playful games, and laughter exercises. Delivered in-person, each session lasted 30-40 minutes and followed a standardized format developed by Dr. Madan Kataria.
  Interventions: Behavioral: Face-to-Face Laughter Yoga Group
- Online Laughter Yoga Group (Experimental): Participants in this group received the same laughter yoga intervention as the face-to-face group, but it was delivered online via Zoom. Sessions were held in the evening hours twice a week over two weeks.This intervention followed the same structure as the face-to-face program, including clapping, breathing, and laughter exercises. Sessions were conducted in real time via Zoom by certified laughter yoga instructors.
  Interventions: Behavioral: Online Laughter Yoga Group

INTERVENTIONS:
Behavioral: Face-to-Face Laughter Yoga Group — In this study, each laughter yoga session lasted approximately 30-40 minutes and consisted of four parts: hand clapping and warm-up exercises, deep breathing exercises, playful games, and laughter exercises. According to Kataria (2011), the first three parts remained consistent across all sessions, while the laughter exercises in the fourth part varied (Kataria 2011). In the first session of each new group, participants were introduced to laughter yoga, its purpose, and objectives, with 10 minutes allocated to this introductory section. As a result, the first session for each group lasted 40 minutes, while the remaining sessions were 30 minutes each. The structure and duration of each session were as follows:
  * Section 1: Hand Clapping and Warm-up Exercises - 5 minutes
  * Section 2: Deep Breathing Exercises - 10 minutes
  * Section 3: Playful Games - 5 minutes
  * Section 4: Laughter Exercises - 10 minutes
  Arms: Face-to-Face Laughter Yoga Group
Behavioral: Online Laughter Yoga Group — In this study, each laughter yoga session lasted approximately 30-40 minutes and consisted of four parts: hand clapping and warm-up exercises, deep breathing exercises, playful games, and laughter exercises. According to Kataria (2011), the first three parts remained consistent across all sessions, while the laughter exercises in the fourth part varied (Kataria 2011). In the first session of each new group, participants were introduced to laughter yoga, its purpose, and objectives, with 10 minutes allocated to this introductory section. As a result, the first session for each group lasted 40 minutes, while the remaining sessions were 30 minutes each. The structure and duration of each session were as follows:
  * Section 1: Hand Clapping and Warm-up Exercises - 5 minutes
  * Section 2: Deep Breathing Exercises - 10 minutes
  * Section 3: Playful Games - 5 minutes
  * Section 4: Laughter Exercises - 10 minutes
  Arms: Online Laughter Yoga Group
Other: control group — Participants in the control group will not receive the laughter yoga intervention. They will continue with their usual daily routines and will only complete pre- and post-test assessments.
  Arms: Control Group

SUMMARY:
The planned study aims to contribute to the existing literature by comparatively evaluating the effects of online and face-to-face laughter yoga interventions on nurses, focusing on stress, sleep quality, and burnout. In line with this purpose, the research hypotheses are as follows:

H1. Laughter yoga intervention provided to nurses has a positive effect on their perceived stress levels.

H2. Laughter yoga intervention provided to nurses has a positive effect on their sleep quality.

H3. Laughter yoga intervention provided to nurses has a positive effect on their burnout levels.

H4. There is a significant difference between the effects of online and face-to-face laughter yoga interventions.

DETAILED DESCRIPTION:
This study investigated whether laughter yoga can help reduce stress, improve sleep, and prevent burnout among nurses. Nurses often work in challenging conditions with long shifts, which can negatively affect their mental and physical health. In this study, nurses were divided into three groups: one received face-to-face laughter yoga, another participated in laughter yoga online, and the third group did not receive any intervention.

Laughter yoga sessions were conducted twice a week for two weeks and included deep breathing, playful activities, and laughter exercises. Participants completed surveys before and after the sessions to measure their stress levels, sleep quality, and signs of burnout.

The results showed that nurses who participated in the online laughter yoga program experienced better sleep, felt less emotionally exhausted, and had a stronger sense of personal accomplishment. These benefits were not observed in the face-to-face or control groups. Interestingly, the program did not significantly reduce stress levels in any of the groups.

This study suggests that online laughter yoga may be a useful and accessible tool to support the well-being of nurses, especially in healthcare settings where in-person wellness programs are difficult to organize.

ELIGIBILITY:
Inclusion Criteria:

* working as a nurse
* over 18 years old

Exclusion Criteria:

* No uncontrolled hypertension
* No history of abdominal surgery in the last three months
* Not suffering from glaucoma, hernia or epilepsy
* Not receiving psychiatric diagnosis and treatment
* Not receiving sleep-related diagnosis and treatment
* having incontinence

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-02-10 (Actual); Study Completion 2025-03-10 (Actual)

PRIMARY OUTCOMES:
Perceived Stress Scale | two week and three week after intervention
  ASQ is designed to measure how stressful some situations in a person's life are perceived. A total score of 0-32 is taken from the scale. It has two subscales: perceived stress (items 1, 2, 3, 7, 8) and perceived coping (items 4, 5, and 6). The scale is evaluated on both total score and subscale scores. A high total score means a high perceived stress level. High scores from the subscales are a negative situation.
Jenkins Sleep Scale | two week and three week after intervention
  It is used in clinical studies to evaluate patients' sleep problems. Patients are asked 4 questions about their sleep problems in the last month and asked to tick the boxes that apply to them. 0 (almost never), 1 (1-3 days per month), 2 (4-7 days per month), 3 (8-14 days per month), 4 (15-21 days per month), 5 (23-31 days per month) It is evaluated as . An increase in the score indicates that the person's sleep quality decreases.
Maslach Burnout Scale | two week and three week after intervention
  This measurement tool consists of a total of 22 items and three subscales. Among these subscales, the emotional exhaustion subscale consists of 9 items, the depersonalization subscale consists of 5 items, and the personal accomplishment subscale consists of a total of 8 items. Scale items are scored as "1: never" and "7: always". It was decided to arrange the scale as a five-degree scale, with the answer options being "0 never" and "4 always". The high level of burnout reflects the high score on the emotional exhaustion and depersonalization subscales and the low score on the personal accomplishment subscale. Moderate levels of burnout reflect moderate scores for all three subscales, while low levels reflect low scores on the emotional exhaustion and depersonalization subscales and high scores on the "personal accomplishment" subscale.

CONTACTS AND LOCATIONS:
Overall Officials: Özge TOPSAKAL, Principal Investigator — Manisa Celal Bayar University
Locations (1):
- Manisa Celal Bayar Üniversitesi Hafsa Sultan Hastanesi, Manisa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No